CLINICAL TRIAL: NCT06189417
Title: Effect Of Health Extension Worker-Led Based Interventions on Improving Self-Management Behavior Among Diabetic Patients in Ethiopia
Acronym: HEWL-SMB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Debre Berhan University (Other)
Collaborators: University of South Africa (Other)
Responsible Party: Principal Investigator, Akine Eshete, Principal Investigator, Debre Berhan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-005/23
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Self-management Behavior and Glycosylated Hemoglobin Levels
Keywords: Health Extension Worker, Self-Management Behavior, Club Based Intervention, People with diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Upon completion of the baseline data collection for both groups, a total of 28 clusters/villages will be selected, each involving a maximum of 20 study participants. These clusters will be evenly distributed, with 14 clusters assigned to the intervention group and 14 clusters allocated to the control group. The HEW-led club-based intervention will be integrated into the health extension package. The intervention will take place once a week during club meetings, lasting approximately 50 minutes for six months. Across all clusters or villages, the intervention group will receive 14 educational sessions within a week.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All clusters of study participants will be geographically isolated, and ensuring that intervention and control groups are not exposed to each other. Study participants, HEW and HDA, will be blinded to the outcome interest of the study to avoid the hawthorn effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A total of 280 study participants are allocated to intervention group
  Interventions: Behavioral: Health Extension Led club based Intervention
- control group (No Intervention): A total of 280 study participants are allocated to control group

INTERVENTIONS:
Behavioral: Health Extension Led club based Intervention — The Health Extension Workers-led club-based intervention primarily focuses on equipping individuals with the necessary knowledge and skills to enhance their self-management behavior. The intervention encompasses education on adopting healthy eating habits, promoting regular exercise, effectively managing weight, and supporting smoking cessation. It emphasizes the importance of regular blood sugar level monitoring, limiting alcohol intake, and reducing sedentary behavior. The intervention also includes counseling to provide guidance and support in adopting and maintaining healthy behaviors. Additionally, it highlights the significance of adhering to medication regimens for optimal health outcomes. If additional medical attention is required, the intervention provides referral services to nearby health facilities.
  Arms: Intervention Group

SUMMARY:
Despite the existence of lifestyle interventions designed to encourage self-management behaviors, the difficulty of adhering to recommended practices remains a widespread issue globally, including in Ethiopia. Traditional approaches to care have demonstrated limited effectiveness in promoting self-management behavior. As a potential solution, a Health Extension Worker-Led club-based intervention has been implemented. Therefore, the aim of this study is to assess the impact of the Health Extension Worker-Led club-based intervention on improving self-management behaviors and glycemic control.

The study will utilize a parallel-group, cluster randomized controlled trial design to investigate its objectives. The main focus of the research is to assess the average increase, both in terms of mean and percentage, in adherence to self-management behaviors and glycemic control. Additionally, the study aims to evaluating the acceptance of the intervention. To evaluate the impact of a Health Extension Worker-led intervention on self-management behavior and levels of glycosylated hemoglobin (HbA1C), a difference-in-difference analysis will be employed. A comparison of the intervention's effects across different groups will be conducted using an independent-sample t-test.

DETAILED DESCRIPTION:
Despite the Ethiopian government's focus on non-communicable diseases, diabetes is increasingly becoming a major public health issue among adults. Unfortunately, diabetes care in numerous countries, including Ethiopia, is inadequate, resulting in undiagnosed cases, low rates of diabetes control, and failure to meet established care standards.

Insufficient readiness of healthcare services, inadequate training of healthcare professionals, and a lack of patient-centered interventions have contributed to inadequate healthcare coverage and suboptimal self-management behavior. The inadequate adherence to self-management behavior has become a critical issue, with half of the patients failing to comply in Ethiopia. Several systematic reviews and meta-analyses consistently indicate that the range for achieving good diabetes self-management behavior is between 49.8% and 51.12%.

To ensure the provision of high-quality diabetes care, it is vital to prioritize patient preferences and needs by adopting a patient-centered approach. The implementation of community-based care programs that prioritize patient-centeredness and aim to enhance patients' understanding of self-care management is of utmost importance. Published evidence strongly indicates that educational interventions can play a significant role in supporting individuals with diabetes to improve their self-care management.

The existing delivery approaches in various countries, including Ethiopia, are insufficient in facilitating the adoption of recommended self-care practices. Therefore, there is an urgent need to implement patient-centered care programs at the community level. To address this issue, a Health Extension Worker-Led club-based intervention has been introduced as a strategic intervention approach to fill this gap. The Health Extension Worker-led club-based intervention is seamlessly integrated into the existing Health Extension Program. The introduction of a community-based intervention has a significant impact on self-management behavior, improves access to chronic disease services, and enhances outcomes for individuals with chronic diseases.

To the best of our knowledge, there is a lack of evidence regarding the impact of a Health Extension Worker-led club based intervention on self-management behaviors in Ethiopia. Therefore, the objective of this study is to assess the impact of the Health Extension Worker (HEW)-led club-based intervention on improving self-management behaviors, glycemic control, and the acceptance of the intervention among individuals with diabetes in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes who have provided informed consent
* Patients with diabetes who do not have any other diabetes-related health complications at the start of the study
* Patients with diabetes who are not pregnant
* Patients with diabetes who have completed six months in the study
* Patients with diabetes who have expressed their intention to remain within the study facility (health post) and community.

Exclusion Criteria:

* Patients who decline to provide consent
* Patients who, based on medical assessment by their physician, are deemed unable to participate in the intervention
* Patients who choose not to continue with the intervention.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean and proportion of diabetic self-management behavior | measured at six months
  The proportion of self-management behaviors will be determined using the Diabetes Self-Care Activity Summary tool. Participants will be requested to report the frequency of these specific behaviors per week using an eight-point Likert scale, ranging from 0 to 7 days. The responses obtained through this scale will be utilized to compute an overall score, with higher average scores indicating greater adherence to self-management behaviors and practices. The study will compare the mean change in self-management behaviors at six months from baseline among the different groups.
Mean and proportion increase in glycemic control | measured at three and six months
  Fasting blood sugar (FBS) and Glycosylated hemoglobin (HbA1C) are widely utilized measures to assess glycemic control. The baseline FBS analysis involves calculating the mean of FBS measurements taken over three consecutive months. During the follow-up period, the analysis is conducted using the mean values of FBS measurements taken over six consecutive months. According to the guideline recommendations of the American Diabetes Association (ADA), glycemic status is considered good if the mean FBS falls between 80 and 130 mg/dL. Glycosylated hemoglobin (HbA1C) levels will be assessed at two time points: three months during follow up and six months after the intervention. The optimal range for glycosylated hemoglobin (HbA1C) levels for individuals with diabetes is below 7% (53 mmol/mol).

SECONDARY OUTCOMES:
Acceptability of a community-based club intervention led by Health Extension Workers | measured at six months
  Acceptability, in this context, refers to the extent to which the intervention is perceived as appropriate, suitable, and desirable by the participating individuals. It assesses the community's willingness to actively engage with and adhere to the intervention, as well as their satisfaction and comfort with the intervention activities and delivery methods. To measure acceptability, participants will be asked to indicate their agreement with a series of statements related to the intervention using a five-point Likert scale, ranging from 1 to 5. The responses obtained through this scale will be utilized to compute an overall score, with higher average scores indicating greater acceptance level. Open-ended questions will also be included to gather participants' perspectives on the intervention content, their experiences with the HEW-led club intervention, and any suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Akine E Abosetugn, MPH, Principal Investigator — Debre Berhan University
Locations (1):
- Debre Berhan University and North Shoa Zone Health Department, Debre Berhan, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MoH., Realizing Universal Health Coverage through Primary Health Care: A Roadmap for Optimizing the Ethiopian Health Extension Program 2020 - 2035. Addis Ababa, Ethiopia: Ministry of Health, 2020. 2020.
- [Background] Bishu K.G, et al., Diabetes in Ethiopia: A systematic review of prevalence, risk factors, complications, and cost. Obesity Medicine, 2019. 15: p. 100132:https://doi.org/10.1016/j.obmed.2019.100132.
- [Background] Zeru MA, Tesfa E, Mitiku AA, Seyoum A, Bokoro TA. Prevalence and risk factors of type-2 diabetes mellitus in Ethiopia: systematic review and meta-analysis. Sci Rep. 2021 Nov 5;11(1):21733. doi: 10.1038/s41598-021-01256-9. PMID 34741064
- [Background] Mulugeta TK, Kassa DH. Readiness of the primary health care units and associated factors for the management of hypertension and type II diabetes mellitus in Sidama, Ethiopia. PeerJ. 2022 Aug 25;10:e13797. doi: 10.7717/peerj.13797. eCollection 2022. PMID 36042860
- [Background] Tesema AG, Peiris D, Abimbola S, Ajisegiri WS, Narasimhan P, Mulugeta A, Joshi R. Community health extension workers' training and supervision in Ethiopia: Exploring impact and implementation challenges for non-communicable disease service delivery. PLOS Glob Public Health. 2022 Nov 9;2(11):e0001160. doi: 10.1371/journal.pgph.0001160. eCollection 2022. PMID 36962619
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2021 Abridged for Primary Care Providers. Clin Diabetes. 2021 Jan;39(1):14-43. doi: 10.2337/cd21-as01. No abstract available. PMID 33551551
- [Background] Dagnew B, Debalkie Demissie G, Abebaw Angaw D. Systematic Review and Meta-Analysis of Good Self-Care Practice among People Living with Type 2 Diabetes Mellitus in Ethiopia: A National Call to Bolster Lifestyle Changes. Evid Based Complement Alternat Med. 2021 Feb 20;2021:8896896. doi: 10.1155/2021/8896896. eCollection 2021. PMID 33688368
- [Background] Ansari R M, et al., Implementation of Chronic Care Model for Diabetes Self-Management: A Quantitative Analysis. Diabetology, 2022. 3(3): p. 407-422.
- [Background] Ketema DB, Leshargie CT, Kibret GD, Assemie MA, Alamneh AA, Kassa GM, Alebel A. Level of self-care practice among diabetic patients in Ethiopia: a systematic review and meta-analysis. BMC Public Health. 2020 Mar 12;20(1):309. doi: 10.1186/s12889-020-8425-2. PMID 32164638
- [Result] FDREMoH, National Strategic Plan for the Prevention And Control Of Major Non-Communicable Diseases, 2013-2017(2020/21-2024/25), Addis Ababa Ethiopia; July 2020. 2020.